CLINICAL TRIAL: NCT03512860
Title: An Open-label, Two-way Cross-over Study to Determine the Effect of Multiple Doses of Valproic Acid on the Pharmacokinetics and Safety of a Single Oral Dose of Estetrol/Drospirenone in Healthy Female Subjects
Brief Title: Estetrol (E4)/Drospirenone (DRSP) Drug-drug Interaction (DDI) Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Estetra (Industry)
Collaborators: Quotient Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: MIT-Es0001-C110; 2017-004280-12 (EudraCT Number)
Record Dates: First submitted 2018-04-19; First posted 2018-05-01 (Actual); Last update posted 2018-12-14 (Actual); Status verified 2018-12

CONDITIONS: Contraception
Keywords: Estetrol; Drospirenone; Uridine diphosphate glucuronosyltransferase-2B7; Drug-drug interaction; Valproic acid
MeSH Terms: interventions — Valproic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- E4/DRSP (Treatment A) - E4/DRSP + VAL (Treatment B) (Experimental): Sequence A-B: A single oral dose of E4 combined with DRSP (Treatment A) will be administered during the Period 1. After a washout, subjects will enter into the Period 2. They will receive the Treatment B which consists in multiple oral doses of VAL for 12 consecutive days and one single oral dose of E4/DRSP on Day 5 of the VAL administration.
  Interventions: Drug: E4/DRSP; Drug: VAL
- E4/DRSP + VAL (Treatment B) - E4/DRSP (Treatment A) (Experimental): Sequence B-A: During Period 1, subjects will receive the Treatment B (multiple oral doses of VAL for 12 consecutive days and one single oral dose of E4/DRSP on Day 5 of the VAL administration) . After a washout, subjects will enter into the Period 2 and receive the Treatment A (a single oral dose of E4 combined with DRSP).
  Interventions: Drug: E4/DRSP; Drug: VAL

INTERVENTIONS:
Drug: E4/DRSP — Administered as specified in the treatment arm.
  Other Names: E4 and DRSP combined tablet
Drug: VAL — Administered as specified in the treatment arm.
  Other Names: Valproic acid; Depakote®

SUMMARY:
The present study is designed to determine the effect of valproic acid (VAL), a UGT2B7 inhibiting drug, on the pharmacokinetics (PK) of estetrol (E4)

DETAILED DESCRIPTION:
In the present study, E4/DRSP will be administered alone (Treatment A) and in combination with VAL (Treatment B) following two sequences A-B or B-A.

ELIGIBILITY:
Inclusion Criteria:

* Healthy premenopausal, aged 18-45 years (inclusive) at the time of signing informed consent.
* For subjects who are sexually active and are of childbearing potential: willing to use a highly effective non-hormonal method of contraception from screening until the follow-up assessment, such as (but not limited to): non-hormonal intra-uterine device (copper IUD), bilateral tubal occlusion, vasectomised partner, or sexual abstinence in a heterosexual relationship; this is acceptable when it is in line with the subject's preferred and usual lifestyle. If a subject is usually not sexually active but becomes active, they, with their partner, must comply with the contraceptive requirements as stated earlier.
* Body weight ≥45 kg, and a body mass index between 18.0 and 30.0 kg/m² (inclusive).
* Negative serum pregnancy test at screening and a negative urine pregnancy test at Day -1.

Exclusion Criteria:

* The use of:

  * any prescription drugs, including oral or vaginal hormonal contraceptives, from 28 days prior to first dose administration until study completion;
  * any herbal medication or dietary supplements acting on cytochrome P450 3A4 (CYP3A4) functions (i.e., St John's Wort), from 28 days prior to first dose administration until study completion;
  * any over-the-counter medication (including paracetamol or dietary supplements (including vitamins and herbal products ), from 14 days prior to first dose administration until study completion. Limited use (i.e., up to 1200 mg/day) of ibuprofen is allowed;
  * any depot progestogen preparations or an injectable hormonal method of contraception, from 6 months prior to the first dose administration until study completion.
* History of hypersensitivity, serious adverse reaction, or existing contraindication to E4, DRSP or VAL, or excipients.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2018-04-12 (Actual); Primary Completion 2018-10-08 (Actual); Study Completion 2018-10-08 (Actual)

PRIMARY OUTCOMES:
Maximum concentration (Cmax) of E4 | 0-168 hr post E4/DRSP dose in both periods 1 and 2 of the two sequences A-B and B-A
  PK sampling
Area under the plasma concentration versus time curve from time 0 to the last determined concentration (AUC0-tdlc) of E4 | 0-168 hr post E4/DRSP dose in both periods 1 and 2 of the two sequences A-B and B-A
  PK sampling
Area under the plasma concentration versus time curve from time 0 to infiny (AUC0-inf) of E4 | 0-168 hr post E4/DRSP dose in both periods 1 and 2 of the two sequences A-B and B-A
  PK sampling

SECONDARY OUTCOMES:
Number of subjects with adverse events as a measure of safety and tolerability | The total study duration (between 50 and 86 days)
Cmax of DRSP | 0-168 hr post E4/DRSP dose in both periods 1 and 2 of the two sequences A-B and B-A
  PK sampling
Cmax of E4-glucuronide metabolites | 0-168 hr post E4/DRSP dose in both periods 1 and 2 of the two sequences A-B and B-A
  PK sampling
AUC0-tdlc of DRSP | 0-168 hr post E4/DRSP dose in both periods 1 and 2 of the two sequences A-B and B-A
  PK sampling
AUC0-tdlc of E4-glucuronide metabolites | 0-168 hr post E4/DRSP dose in both periods 1 and 2 of the two sequences A-B and B-A
  PK sampling
AUC0-inf of DRSP | 0-168 hr post E4/DRSP dose in both periods 1 and 2 of the two sequences A-B and B-A
  PK sampling
AUC0-inf of E4-glucuronide metabolites | 0-168 hr post E4/DRSP dose in both periods 1 and 2 of the two sequences A-B and B-A
  PK sampling

CONTACTS AND LOCATIONS:
Overall Officials: Sharan Sidhu, Principal Investigator — Quotient Sciences
Locations (1):
- Quotient Sciences, Ruddington, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided